CLINICAL TRIAL: NCT06745232
Title: The Use of a New Stereophotogrammetry System to Capture Intra-operative Complete-arch Impression
Brief Title: New Stereophotogrammetry System to Capture Complete-arch Impression
Status: Recruiting | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Paolo Carosi, Post-doc Researcher, University of Rome Tor Vergata
Other Study IDs: FASTMAPPROSPECTIVE
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Prosthetic Complication; Prosthesis Failure, Dental
Keywords: fixed prosthesis; stereophotogrammetry; immediate loading
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- FAST MAP: Patients with complete arch restorations loaded immediately with a full digital workflow using stereophotogrammetry Intraoral impression
  Interventions: Device: FAST MAP

INTERVENTIONS:
Device: FAST MAP — Patients with complete arch restorations loaded immediately with a full digital workflow using stereophotogrammetry Intraoral impression

SUMMARY:
Patients in need of complete arch restorations will be treated with dynamic navigation system. Once the implants are positioned, a new system of stereophotogrammetry will record the implant positions to capture a precise impression to deliver a fixed screw retained interim prosthesis

ELIGIBILITY:
Inclusion Criteria:

1. Healthy patients aged ≥18 years
2. Full mouth bleeding and full mouth plaque index lower than or equal to 25%
3. Bone height for at least 10 mm long implants
4. Bone width of at least 5 mm and 6 mm for narrow (NP 3.75/3.5 mm) and regular (RP 4.3 mm) implants, respectively
5. Fresh extraction sockets with an intact buccal wall
6. At least 4 and 5 mm of bone beyond the root apex in the mandible and maxilla
7. Minimal insertion torque of 45 Ncm

Exclusion Criteria:

1. General medical (American Society of Anesthesiologists, ASA, class III or IV) and/or psychiatric contraindications
2. Pregnancy and/or breastfeeding
3. Any interfering medication such as steroid therapy or bisphosphonate therapy
4. Alcohol and/or drug abuse
5. Heavy smoking (>10 cigarettes/day)
6. Radiation therapy to head or neck region within 5 years
7. Untreated periodontitis
8. Acute and chronic infections of the adjacent tissues or natural dentition
9. Severe maxillomandibular skeletal discrepancy
10. High and moderate parafunctional activity
11. Absence of opposite teeth

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients in need of complete arch rehabilitations with dental implants and fixed dental prosthesis
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Prosthetic Success | 3 months
  Prosthetic success of interim prosthesis in term of passivity and tissues adaptability

CONTACTS AND LOCATIONS:
Locations (1):
- PTV, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No